CLINICAL TRIAL: NCT04538729
Title: Use of Alternative Therapy in Acne Vulgaris Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Melek Aslan Kayıran, M.D., Istanbul Medeniyet University
Other Study IDs: IstanbulMU9
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Acne Vulgaris — Alternative medicine and complementary therapies that acne vulgaris patients apply without informing the doctor, how they learn these techniques, what make them use these techniques for their illness

SUMMARY:
Acne Vulgaris is a chronic skin disease. However, chronic and repetitive due to the quality of life and psychological status of patients can affect. Today, although the treatment is repetitive, chronic and requires follow-up due to the disease patients can turn to alternative and complementary medicine techniques. In recent years, studies on alternative medicine and complementary therapies have been noted in the medical literature. These studies also include Case Reports related to acne vulgaris. However, in our country, there is no study that tells us whether patients with acne vulgaris apply these treatments or not and what the practitioners think about the success of the treatment. The aim of the study will be to clarify issues such as whether patients with Acne Vulgaris apply alternative medicine and complementary therapies for their disease.

ELIGIBILITY:
Inclusion Criteria:

* Acne vulgaris Patients between age 12-60

Exclusion Criteria:

* the ones who don't want to answer the questions

Ages: 12 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Acne vulgaris Patients between age 12-60
Sampling Method: Probability Sample
Enrollment: 1571 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
acne vulgaris questionnaire | september 2020
  Alternative medicine and complementary therapies that acne vulgaris patients apply without informing the doctor, how they learn these techniques, what make them use these techniques for their illness

CONTACTS AND LOCATIONS:
Locations (1):
- Melek Aslan Kayıran, Istanbul, Turkey (Türkiye)